CLINICAL TRIAL: NCT06914349
Title: Antecolic Versus Retrocolic Gastrojejunostomy Following Pancreaticoduodenectomy: a Prospective Randomised Study
Brief Title: Antecolic Versus Retrocolic Gastrojejunostomy During Whipple's Procedure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Chrysoula-Christina Kolla, MD, Msc, University of Thessaly
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: University hospital of Larissa
Record Dates: First submitted 2025-03-30; First posted 2025-04-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Cancer Resectable; Pancreas Neoplasms
Keywords: Gastrojejunostomy; Whipple's; Antecolic; Retrocolic
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antecolic gastrojejunostomy (Active Comparator)
  Interventions: Procedure: Antecolic gastrojejunostomy
- Retrocolic gastrojejunostomy (Active Comparator)
  Interventions: Procedure: Retrocolic gastrojejunostomy

INTERVENTIONS:
Procedure: Antecolic gastrojejunostomy — Gastrojejunostomy in front of the transverse colon
  Arms: Antecolic gastrojejunostomy
Procedure: Retrocolic gastrojejunostomy — Gastrojejunostomy through the transverse mesocolon
  Arms: Retrocolic gastrojejunostomy

SUMMARY:
Aim: This randomized clinical study aims to compare occurrence of DGE in patients undergoing either antecolic or retrocolic gastrojejunostomy following pancreaticoduodenectomy.

Methods: Participants of this study will be patients undergoing pylorus preserving pancreaticoduodenectomy at the Surgical Department of the University Hospital of Larissa. Patients will be randomized to undergo either an antecolic or a retrocolic gastrojejunostomy and the occurrence of DGE will then be compared between the two groups. Individuals younger than 18 or older than 75 years old, as well as patients who do not consent to participate in this trial, will be excluded.

Expected results: Based on available literature, antecolic gastrojejunostomy may be related with a lower incidence of DGE, without a statistically significant difference between the two methods. We aim to show if one of the two methods of gastrointestinal reconstruction (antecolic versus retrocolic) affects DGE.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* Elective pancreaticoduodenectomy
* Signed consent form

Exclusion Criteria:

* Age under 18 years old
* Patients who are participants in other trials that may affect the results of this study
* Patients who do not consent to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-03-30 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Delayed Gastric Emptying | 3 years
  The occurence of delayed gastric emptying will be compared between two groups of patients: those who undergo an antecolic gastrojejunostomy and those who undergo a retrocolic approach.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Symeonidis, Study Chair — University of Thessaly
Locations (1):
- University of Thessaly, Larissa, Greece

IPD SHARING:
Plan to Share IPD: Undecided